CLINICAL TRIAL: NCT06242366
Title: Effects of Transitional Care Program in Stroke Patients on Self-care Behavior, Quality of Life, and Hospital Readmission: A Randomized Controlled Trial.
Brief Title: Transitional Care Program in Stroke Patients With Hemiplegia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA. MURA2023/337; U034hh/66 (Other: BMA Human Research Ethics Committee.)
Record Dates: First submitted 2024-01-24; First posted 2024-02-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke; Transitional Care; Hemiplegia
Keywords: Quality Of Life; Self-care behavior; Hospital Readmission; Transitional care; Stroke patients
MeSH Terms: conditions — Ischemic Stroke; Hemiplegia

STUDY DESIGN:
Intervention Model Description: This study based on Transitional Care Model by Naylor. Sixty participants with stroke patients with hemiplegia and can use Line Application will be recruited. These participants are stratified block randomization using NIHSS (5-9) and (10-14) score 30 participant each and then sample random into 2 groups; control group (n=30) and intervention groups (n=30).
  The program consisted of 2 phases: 1) Phases I during hospital admission and 2) Phases II following hospital discharge for 12 weeks will collecting the data are 1) The Personal Data Form, 2) The Self-care Behavior Questionare and 3) The Stroke Impact Scale (SIS) 3.0. Data will be analyzed using descriptive statistics and two-way repeated measures ANOVA.
Who Masked: Participant, Outcomes Assessor
Masking Description: These Sixty participants are stratified block randomization using NIHSS (5-9) and (10-14) score 30 participant each and then sample random into 2 groups; control group (n=30) and intervention groups (n=30) by Investigator . they do not know that their group.
  The Outcomes Assessor will be collecting the data for primary and secondary outcome for 4 and 12 weeks and do not who are control or intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In this arm, the participant will receive standard nursing care and the program from an investigator.
  The program consisted of 2 phases: 1) Phases I during hospital admission when they are stable will receive a program total 4 times for education about stroke, self-care, rehabilitation, and complication prevention and
  2) Phases II following hospital discharge within 24 hours then every 1 week until 4 weeks by Line Application visit. following self-care management, find limit to their self-care.
  and Outcomes Assessor will visit to collect data 3 times
  1. In-hospital period
  2. after hospital discharge 4 weeks
  3. after hospital discharge 12 weeks
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): In this arm, the participant will receive only standard nursing care. and Outcomes Assessor will visit to collect data 3 times
  1. In-hospital period
  2. after hospital discharge 4 weeks
  3. after hospital discharge 12 weeks

INTERVENTIONS:
Behavioral: Intervention group — Intervention 2 phases Phases 1) In-hospital period (4 times and 30-60 mins/times) intervention includes Stroke education, Rehabilitation, environmental management, and complication prevention. Intervention participants will receive a booklet (choose between hard copy or electronic copy) self-care for stroke patients, Rehabilitation clip, and Self-care record form.
  Phases 2) after hospital discharge 5 times (first times within 24 hours after hospital discharge) and (second-fifth time: 1 time/weekly)15-30 mins/times by Line Application for repeat and following education, rehabilitation complication prevention and finding limit to self-care management.
  Arms: Intervention group

SUMMARY:
This study examines the effects of a transitional care program in stroke patients on self-care behavior, quality of life, and hospital readmission.

The research conceptual framework is based on the Transitional Care Model by Naylor. Sixty participants with stroke patients at Charoenkrung Pracharak Hospital will be recruited. These participants are stratified by block randomization using NIHSS score and divided into 2 groups; a control group (n=30) and an intervention group (n=30).

The program consisted of 2 phases: 1) Phase I during hospital admission and 2) Phase II following hospital discharge

DETAILED DESCRIPTION:
This study is to examine the effects of a transitional care program in stroke patients on self-care behavior, quality of life, and hospital readmission.

The research conceptual framework base on Transitional Care Model by Naylor. Sixty participants with stroke patients at Charoenkrung Pracharak Hospital will be recruited. These participants are stratified block randomization using NIHSS score and divide into 2 groups; control group (n=30) and intervention groups (n=30).

The program consisted of 2 phases: 1) Phases I during hospital admission and 2) Phases II following hospital discharge for 4 weeks. The instruments used in this study for collecting the data are 1) The Personal Data Form, 2) The Self-care Behavior Questionare and 3) The Stroke Impact Scale (SIS) 3.0. Data will be analyzed using descriptive statistics and two-way repeated measures ANOVA.

The result of this study will be used to develop guideline for nursing care in stroke patients during the transition from hospital to home. This program will help the patients improve their self-care, quality of life, and reduce hospital readmission

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years old.
* The first diagnosis is acute ischemic stroke.
* Hemiplegia
* NIHSS 5-14 point (moderate impairment)
* Telephone and Line Application used.
* Can read and communicate in Thai language
* Accept participants to research and inform consent.

Exclusion Criteria:

* Aphasia
* The Six Item Cognitive Impairment Test: 6CIT from 8 points in age from 60 years old.
* Participants with illness severity or dead during the study.
* Reject the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Compare Mean differences of Quality Of Life on stroke patient. | Baseline, 4 weeks, 12 weeks
  Each participant was asked using by The Stroke Impact Scale: SIS 3.0 develop by Duncan, Bode, Lai, & Perera, 2003 (Thai version by Garnjanagoonchorn A, and Dajpratham P, 2015) is a 59-item self-report assessment of stroke outcome used to assess HRQoL. There are 8 domains: strength, hand function, mobility, physical and instrumental activities of daily living, memory and thinking, communication, emotion, and social participation. Each item is rated using a 5-point Likert scale. The patient rates his/her difficulty completing each item, where: 1 = an inability to complete the item, 5 = no difficulty experienced at all. An extra question on stroke recovery asks that the client rate on a scale from 0 - 100 how much the client feels that he/she has recovered from his/her stroke. Scores for each domain range from 0 to 100; 0 = no recovery, 100 = full recovery. and higher scores indicate a better HRQoL. will use two-way repeated-measures ANOVA statistics for data analysis.
Compare Mean differences of self-care behavior on stroke patient. | Baseline, 4 weeks, 12 weeks
  Each participant was asked using by self-care behavior questionnaire (Thai version) develop by Kasama Chiangtong (2011) is a 15-item self-report assessment of self-care behavior. Each item is rated using a 4-point Likert scale, where: 0 = never, 1= sometimes (1-2 times/week), 2= often (3-5 times/week), 3= regular. Scores range from 11 to 45 and higher scores indicate a high self-care behavior management. will use two-way repeated-measures ANOVA statistics for data analysis.

SECONDARY OUTCOMES:
Number of Participants with Hospital Readmission. | 4 weeks.
  Each participants were monitored for up to 4 weeks after hospital discharge. This is the number of participants who have had ischemic stroke with readmission within 28 days after hospital discharge with recurrence of the disease or complications from stroke. rate of Hospital Readmission will use descriptive statistics for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rungnapa Premkamol, Principal Investigator — Mahidol University
Locations (1):
- Charoenkrung Pracharak Hospital, Bang Kho Laem, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional care of older adults hospitalized with heart failure: a randomized, controlled trial. J Am Geriatr Soc. 2004 May;52(5):675-84. doi: 10.1111/j.1532-5415.2004.52202.x. PMID 15086645
- [Result] Wong FK, Yeung SM. Effects of a 4-week transitional care programme for discharged stroke survivors in Hong Kong: a randomised controlled trial. Health Soc Care Community. 2015 Nov;23(6):619-31. doi: 10.1111/hsc.12177. Epub 2014 Dec 3. PMID 25470529
- [Result] Suphimol P. The Effect of Healtth Education Program for Hypertension Prevention Among Risk Group Aged 35-59 Years in Songdao District Of Sakonnakhon Province.: Konkaen University; 2009. (In Thai)